CLINICAL TRIAL: NCT01403246
Title: Phase I-II Multicenter Study to Assess the Efficacy and Safety of the Chlorambucil + Lenalidomide Combination and Lenalidomide Maintenance Therapy in Untreated Elderly Pts With CLL. EudraCT Number 2009-013415-35
Brief Title: Chlorambucil + Lenalidomide and Lenalidomide Maintenance in Untreated Elderly With Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow patient enrollment and new molecules for chronic lymphoid leukemia, have importantly reduced the interest of conducting the phase II of this study.
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLL0709
Record Dates: First submitted 2011-01-13; First posted 2011-07-27 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Lenalidomide; Chlorambucil; No previous treatment
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide with Chlorambucil (Experimental)
  Interventions: Drug: Lenalidomide; Chlorambucil

INTERVENTIONS:
Drug: Lenalidomide; Chlorambucil — MTD of lenalidomide given in combination with chlorambucil

SUMMARY:
This is a phase I multicenter, open label study in previously untreated and elderly patients (> 60 years) with CLL: a non-comparative phase aimed at defining the MTD of lenalidomide given in combination with chlorambucil and the efficacy and safety of the lenalidomide and chlorambucil combination.

DETAILED DESCRIPTION:
All patients will receive six monthly courses of the chlorambucil (C) and lenalidomide (L) schedule consisting of 8 days of C (d1-d8) combined with L given daily until response assessment which will take place 12 weeks from the start (d+1) of course VI, while patients continue their treatment with lenalidomide daily.

In the first phase of the induction phase of the study the dose of L given with C will be gradually escalated to reach the MTD.

Patients who will achieve a response after 6 courses of CL induction phase -PR, CRi, CR

The study was first designed to be a phase I-II trial, yet the second phase of the study was not conducted due to different reasons, among which: poor accrual and lack of interest.

ELIGIBILITY:
Inclusion Criteria:

* CLL diagnosis according to the 2008 revised NCI criteria.
* Age > 65 years or between 60 and 65 years if not suitable for fludarabine-based regimens according to the investigator's judgment.
* ECOG performance status of ≤2 at study entry.
* No previous treatment.
* Advanced stage or progressive CLL according to the 2008 revised NCI criteria.
* Disease-free of prior malignancies other than CLL for ≥3 years, with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Able to take low molecular weight heparin or in alternative, low-fixed-dose warfarin or, in alternative, low-dose aspirin.
* Able to adhere to the study visit schedule and other protocol requirements.
* Female subjects of childbearing potential(FCBP) must:

  * Understands the potential teratogenic risk to the unborn child and the need for effective contraception;
  * Be capable of complying with effective contraceptive measures.
  * Be informed and understand the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy.
  * Understand the need to commence the study treatment as soon as study drug is dispensed following a negative pregnancy test.
  * Uderstand the need and accepts to undergo pregnancy testing based on the frequency outlined in this protocol.
  * Contraception.
  * Females of childbearing potential (FCBP) enrolled in this protocol must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 28 days after study treatment discontinuation.
  * The two methods of reliable contraception must include one highly effective method and one additional effective (barrier) method. FCBP must be referred to a qualified provider of contraceptive methods if needed. The following are examples of highly effective and additional effective methods of contraception:
  * Highly effective methods:

    1. Intrauterine device (IUD)
    2. Hormonal (birth control pills, injections, implants)
    3. Tubal ligation
    4. Partner's vasectomy
  * Additional effective methods:

    1. Male condom
    2. Diaphragm
    3. Cervical Cap
* Because of the increased risk of venous thromboembolism in patients with multiple myeloma taking lenalidomide and dexamethasone, combined oral contraceptive pills are not recommended. If a patient is currently using combined oral contraception the patient should switch to one of the effective method listed above. The risk of venous thromboembolism continues for 4 to 6 weeks after discontinuing combined oral contraception. The efficacy of contraceptive steroids may be reduced during co-treatment with dexamethasone.
* Implants and levonorgestrel-releasing intrauterine systems are associated with an increased risk of infection at the time of insertion and irregular vaginal bleeding. Prophylactic antibiotics should be considered particularly in patients with neutropenia.
* Pregnancy testing.
* FCBP must have two negative pregnancy tests prior to starting study drug. The first pregnancy test must be performed within 10 to 14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug.
* FCBP must agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
* Females must agree to abstain from breastfeeding during study participation and for at least 28 days after study drug discontinuation.
* Male patients must:

  * Understand the potential teratogenic risk if engaged in sexual activity with a pregnant female or a female of childbearing potential.
  * Must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.
  * If pregnancy or a positive pregnancy test does occur in the partner of a male study patient during study participation, the investigator must be notified immediately.
* Female and male patients:

  * should be instructed never to give this medicinal product to another person and to return any unused capsules to the study doctor at the end of treatment.
  * Should not donate blood during therapy and for at least 28 days following discontinuation of study drug.
  * Male patients should not donate blood, semen or sperm during therapy or for at least 28 days following discontinuation of study drug.
* Laboratory test results within these ranges:

  * Serum creatinine ≤1.5 mg/dL and creatinine clearance ≥ 60mL/min
  * Total bilirubin ≤1.5 mg/dL
* AST (SGOT) and ALT (SGPT) ≤1.5 x ULN.
* All patients must be able to understand and voluntarily sign the informed consent form.

Exclusion criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* A CIRS score > 6.
* Pregnant or Lactating Females.
* Known positive serology for HIV or active hepatitis B or C.
* Active infection requiring systemic anti-viral, antibiotic or anti-fungal therapy.
* History of tuberculosis within the last five years or recent exposure to tuberculosis equal to or less than 6 months.
* History of renal failure requiring dialysis.
* Known presence of alcohol and/or drug abuse.
* History of thrombosis, thromboembolism within one year.
* Hearth failure, arrhythmia.
* ≥ grade 2 neuropathy.
* Uncontrolled hyperthyroidism or hypothyroidism.
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
* One or more laboratory abnormalities:
* calculated creatinine clearance (Cockroft-Gault) <60mL/min;
* electrolyte abnormalities according to the Cairo Bishop definition of laboratory TLS.
* GOT, GPT, γGT > 1.5 x upper limit of normal value;
* serum bilirubin >1.5 mg/dL.
* Lactose Intolerance.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foà, Principal Investigator — Umberto I - Dipartimento di Biotecnologie Cellulari ed Ematologia Cellulari; Francesca Romana Mauro, Co-Coordinator, Principal Investigator — Umberto I - Dipartimento di Biotecnologie Cellulari ed Ematologia
Locations (10):
- Italy (10):
  - Azienda Spedali Civili, Brescia
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Clinica Ematologica - Università degli Studi, Genova
  - UO Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Umberto I di Roma - Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - SS.C. di Oncoematologia - Dipartimento di Medicina Clinica e Sperimentale - Azienda Ospedaliera - S. Maria Di Terni, Terni

REFERENCES:
- See also: GIMEMA Foundation Webpage — http://www.gimema.it

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide and Chlorambucil
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 9
Age, Customized [Mean (Full Range); unit: years] | 72 [67 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  Italy | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxic Events (DLT) of Lenalidomide Given in Combination With Chlorambucil.
Time Frame: At maximum 8 months from induction therapy start
Measure: Number; unit: Toxic events
Arm/Group | Study Group
Number analyzed (Participants) | 9
Toxic events | 0

ADVERSE EVENTS:
Time Frame: 3 years and 3 months
Description: The adverse events in the present study report have been classified according to the CTCAE grading. These are included under the Serious Adverse Events, although the fields in the form do not allow to specify grading.
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=9)
Neutropenia (Blood and lymphatic system disorders) | 2 (5)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs of participating centres may disclose their centre's results only after the main study publication has been released, so that a single centre experience can be compared to the study overall results and give a more appropriate view of the study.